CLINICAL TRIAL: NCT07220967
Title: A Randomized Controlled Trial to Determine the Efficacy of Local Antibiotic Delivery in the Prevention of Breast Tissue Expander-Associated Infections
Brief Title: A Study of Antibiotic Delivery to Prevent Infection After Breast Tissue Expander Placement
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-278
Record Dates: First submitted 2025-10-22; First posted 2025-10-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: Breast Tissue Expander Placement; Stimulan Rapid Cure; Local Antibiotic Delivery; Prevent Infection; 25-278
MeSH Terms: conditions — Breast Neoplasms | interventions — Tissue Expansion Devices; Vancomycin; Gentamicins

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled study to compare the outcomes of immediate tissue expander (TE)-based breast reconstruction with and without antibiotic beads.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients randomized to Tissue Expander (TE) + antibiotic beads (Experimental)
  Interventions: Procedure: Tissue Expander (TE); Drug: Vancomycin and Gentamicin; Device: Stimulan Rapid Cure
- Patients randomized to Tissue Expander (TE) only (Active Comparator)
  Interventions: Procedure: Tissue Expander (TE)

INTERVENTIONS:
Procedure: Tissue Expander (TE) — Tissue Expander (TE)
Drug: Vancomycin and Gentamicin — Given through Stimulan Rapid Cure during surgery
  Arms: Patients randomized to Tissue Expander (TE) + antibiotic beads
Device: Stimulan Rapid Cure — Vancomycin and Gentamicin given through Stimulan Rapid Cure during surgery
  Arms: Patients randomized to Tissue Expander (TE) + antibiotic beads

SUMMARY:
The researchers are doing this study to find out whether Stimulan Rapid Cure works to reduce the risk of infections in people getting tissue expanders placed during mastectomy. The researchers will also study whether Stimulan Rapid Cure affects the risk of seroma, a possible complication of surgery that involves fluid buildup under the skin.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Aged 18 years or older
* Planned to undergo mastectomy for breast cancer, genetic predisposition to and/or strong family history of breast cancer, or other prophylactic indication
* Planned to undergo unilateral or bilateral immediate breast reconstruction (i.e., reconstruction at the time of mastectomy) with prepectoral TE placement at MSK
* BMI less than 40 kg/m2
* Not actively smoking or using other nicotine products within 6 weeks of surgery
* No contraindications to Stimulan antibiotic bead placement: hypercalcemia, severe vascular or neurological disease, uncontrolled diabetes, pregnancy, and severe degenerative bone disease
* No known allergy to calcium sulfate, vancomycin, or gentamicin
* No impaired decision-making capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 392 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Surgical site infections (SSI) incidence | within 90 days postoperatively
  We will define SSI as clinically evident local signs or symptoms of infection (e.g., breast erythema, swelling, and/or warmth without an alternative etiology [seroma, radiation]; purulent drainage; aspirate with positive cultures), with or without systemic signs or symptoms (e.g., fever, leukocytosis), that occur within 90 days postoperatively

SECONDARY OUTCOMES:
Compare the rates of seroma | within 90 days postoperatively
  Seroma is defined as >50 cc of periprosthetic fluid that is aspirated during tissue expansions or otherwise drained (e.g., by Interventional Radiology). Seroma will be assessed at the patient level such that unilateral or bilateral seroma in a patient will be considered a single seroma event for the purposes of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Rochlin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/